CLINICAL TRIAL: NCT03908762
Title: Use of a Digital Therapeutic and Connected Devices to Support Insulin Titration
Brief Title: mHealth Titration and Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amalgam Rx, Inc. (Industry)
Collaborators: Kansas City Area Life Sciences Institute, Inc. (Other); University of Kansas (Other); LifeScan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00142758
Record Dates: First submitted 2019-04-08; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Complication
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications | interventions — Magnets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iSage (Experimental): The provider will choose a treatment algorithm embedded within the app and set the parameters to make insulin dose adjustments no less frequently than every 7 days. The app is downloaded by the patient while in the examination room, and the patient is instructed to perform daily fasting glucose fingerstick measurements and follow the app's recommendations for insulin adjustment. Data on telephone or visit contact with a healthcare provider will be collected via the EMR. Hypoglycemic events (defined as blood glucose <70 mg/dl, measured or perceived) are recorded in the iSage application as well as patient report. Providers are asked to review the patients transmitted blood sugar logs as necessary, and those reviews are recorded. Return visits are managed by the HCP and will be logged as resource utilization.
  Interventions: Device: iSage App with connected glucometer
- Conventional Management (Active Comparator): Our clinic uses a modified treat-to-target algorithm which is summarized on a 3 x 5 refrigerator magnet. In the case of glargine or detemir (Basaglar, Lantus, Levemir) adjustments of 1 unit of insulin/day are made until the fasting blood sugars (2 of 3 consecutive values) are 80-130 mg/dl. In the instance of Toujeo or Tresiba, adjustments of 2 units are made every 5 days. Volunteers will have meters downloaded (or interviewed where necessary) to obtain data on fasting blood sugar and episodes of hypoglycemia (perceived or measured <70 mg/dl). The PCP is free to request glucose logs and set return appointments as needed to manage the patient.
  Interventions: Behavioral: Magnet

INTERVENTIONS:
Device: iSage App with connected glucometer — Providers prescribe an insulin dosing plan to patients and provide them with a connected glucometer. The patient's plan is administered through a mobile application. In addition, patients receive education and guidance on insulin administration.
  Arms: iSage
Behavioral: Magnet — Patients are given a refrigerator magnet with an insulin titration algorithm and are asked to follow the instructions on the magnet.
  Arms: Conventional Management

SUMMARY:
The principal objective of this application is to improve glycemic control of diabetic patients treated with basal insulin through use of an innovative, FDA-cleared smartphone-based insulin titration application connected to Bluetooth enabled glucose meters. iSage Rx (isageapp.com) allows providers to prescribe basal insulin treatment plans to patients and manages basal insulin doses utilizing clinically proven algorithms. In this pilot study, we hypothesize that this user-friendly application and seamless data capture will improve glycemic control (achieve HgbA1c <7%) and reduce the frequency and severity of hypoglycemia. Exploratory measures will include healthcare resource utilization and patient and provider satisfaction. The basal insulin titration algorithms used in iSage have had thousands of user-years' experience in FDA-mandated, closely supervised clinical trials, both for long-acting insulins (e.g., Lantus, Levemir) that have been available for a long time and for the newer ultra-long-acting ones (e.g., Tresiba, Toujeo). However, the effectiveness of iSage with a connected glucose meter has not been studied in a "real world" clinical environment. Broad use of such an application and connected devices will, we believe, prove to be cost-effective, favor early and appropriate prescription of insulin, reduce provider effort, shorten time to achieve glycemic goals, and simplify the transition to basal insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* T2DM (WHO criteria) treated with basal insulin (glargine, detemir, degludec)
* HgbA1c 8 or above
* GFR >60 ml/min within the last 12 months
* English speaking, informed consent
* Has an Android or iOS based compatible smartphone (iOS 9.0 or above; Android 4.4 or above)
* Currently performs at least 3 fasting fingerstick glucose measurements/week
* Have a PCP within the KU Health System

Exclusion Criteria:

* Diagnosis of hypoglycemic unawareness within 6 months of enrollment
* Diagnosis of hyperglycemic hyperosmolar non-ketotic coma (HONK) or diabetic ketoacidosis (DKA) within 6 months of enrollment
* Recent (within the last 6 months)/current use of non-topical steroids
* Insulin requirements in excess of 1U/kg per day
* Use of pioglitazone or another thiazolidinedione (TZD)
* In the opinion of the provider, HgbA1c goals should adjusted above 7% due to infirmity, unstable cardiovascular disease, etc.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in A1C | 3 Months
  Mean and Median Change from Baseline

SECONDARY OUTCOMES:
A1C in Target | Baseline to 3 months
  Percentage of patients with an A1C < 7
Rate of Hypoglycemia | Baseline to 3 months
  Percentage of glucose readings <70

CONTACTS AND LOCATIONS:
Locations (1):
- Cray Diabetes Self-Management Center, Kansas City, Kansas, United States